CLINICAL TRIAL: NCT03329365
Title: Paroxysmal Nocturnal Hemoglobinuria and Embolic Strokes of Undetermined Source (ESUS) and Transient Ischemic Attacks of Undetermined Source (ETUS)
Brief Title: Paroxysmal Nocturnal Hemoglobinuria in ESUS & ETUS
Status: Active, not recruiting | Type: Observational
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HSREB109061
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-03

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria; Embolic Stroke of Undetermined Source; Transient Ischemic Attack; Cerebral Vein Thrombosis
Keywords: Flow cytometry; Lactate dehydrogenase (LDH) release; Anemia; Cytopenia
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Ischemic Attack, Transient; Intracranial Thrombosis; Anemia; Cytopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- ESUS/ETUS: Patients with embolic ischemic stroke or transient ischemic attack of undetermined source
- SSS-CVTUS: Patients with superior sagittal sinus cerebral venous thrombosis of undetermined source

SUMMARY:
Paroxysmal nocturnal hemoglobinuria (PNH) is a rare acquired clonal hematological disorder, which can cause arterial or venous thrombosis. The frequency of PNH in young patients (< 50 years old) with embolic stroke (ESUS), transient ischemic attack (ETUS) or superior sagittal sinus cerebral venous thrombosis (SSS-CVTUS) of undetermined source, is currently unknown. This study proposes to recruit ESUS, ETUS, SSS-CVTUS patients to determine the frequency of PNH diagnosis confirmed by flow cytometry in these patient populations.

DETAILED DESCRIPTION:
Paroxysmal nocturnal hemoglobinuria (PNH) is a rare acquired clonal hematological disorder leading to red blood cells hemolysis and thrombosis. PNH has been reported to be the cause of cerebral venous thrombosis and embolic ischemic strokes and is sometimes diagnosed after the ischemic event. In young patients with embolic ischemic stroke of undetermined source (ESUS), thrombophilia is usually investigated. However, access to PNH testing is limited. PNH is rarely investigated in stroke patients and its contribution to the pathophysiology of ESUS is unknown. The investigators hypothesize that this condition is underdiagnosed, resulting in potential preventive opportunities being lost, since PNH can be successfully treated.

This observational study aims to determine the frequency of PNH among young (≤50 years old) patients with recent ESUS or embolic transient ischemic attacks (TIA) of undetermined source (ETUS) and patients with SSS-CVT of undetermined source (SSS-CVTUS).

Patients with ESUS or ETUS will be first screened for: (a) evidence of hemolysis based on their plasma lactate dehydrogenase (LDH) levels, (b) unexplained anemia based on their hemoglobin (Hb) levels, and (c) unexplained cytopenia (e.g., neutropenia and thrombocytopenia). Flow cytometry analysis for PNH will be performed with blood samples collected from subjects with abnormal level of plasma LDH (1.5X ULN) or unexplained anemia or cytopenia.

Patients with SSS-CVTUS will undergo flow cytometry without prior screening.

In addition, plasma and DNA samples will be collected in an optional sub-study for future analysis of DNA mutations related to specific PNH phenotypes in patients with stroke.

ELIGIBILITY:
Inclusion Criteria:

General:

* Participants with embolic ischemic stroke (ESUS), embolic transient ischemic attack (ETUS) or cerebral venous thrombosis (CVTUS) of undetermined source.

For transient ischemic attack (TIA):

One of the following criteria needs to be fulfilled to be considered as embolic TIA:

* Focal symptoms suggesting involvement of de cerebral cortex in the middle cerebral artery (MCA) territory (e.g., aphasia, neglect, apraxia, dystextia, anosognosia, isolated leg, arm or hand weakness). Some of these symptoms have been described as associated with subcortical fibers connecting cortical areas as well but, despite this, they are usually related to cortical localizations. Patients with hemianopia will be included only if hemianopia is not the primary symptom or an isolated symptom.
* Rapidly resolving hemispheric symptoms. This concept comprises two components: (a) sudden onset hemispheric syndrome: sudden onset of symptoms and signs implicating extensive ischemia in the internal carotid artery (ICA) or MCA territories, including hemiparesis, hemianopia, conjugate eye deviation, other cortical signs, or altered consciousness; and (b) spectacular shrinking deficit: improvement within 24 hours (approximately).
* Symptoms involving more than one vascular territory within a single hemisphere (e.g. left sided weakness + left homonymous hemianopia) or both (e.g., left sided weakness and aphasia in a right-handed patient).
* Simultaneous embolization to other organs (e.g., bowel, spleen, liver, kidneys, toes).
* Transient monocular blindness (amaurosis fugax) with no evidence of giant cell arteritis (e.g., normal erythrocyte sedimentation rate).
* No definite cortical symptoms but neuroimaging evidence of prior (chronic) typical infarct (wedge shaped, involving the cerebral cortex).

All of the following criteria must be fulfilled to be considered as TIA of undetermined source:

* No neuroimaging evidence of an acute brain infarct within the brain region(s) responsible for the presenting symptoms.
* Absence of extracranial or intracranial atherosclerosis causing ≥50% luminal stenosis in arteries supplying the area of ischemia.
* No major-risk cardioembolic source of embolism.
* No other specific cause of stroke identified (e.g., arteritis, dissection, migraine, vasospasm, or drug abuse).
* No persistent neurological focal symptoms at the time of neurological examination. The presence of persistent neurological focal symptoms in the absence of a visible brain infarct on DWI MRI will be regarded as a "clinically confirmed stroke with negative DWI MRI".

Exclusion Criteria:

General:

* Inability to provide informed consent

For stroke patients:

* Evidence of >50% stenosis of the internal carotid artery (ICA) or MCA ipsilateral to the qualifying ischemic stroke on neurovascular imaging studies.
* Ischemic stroke involving deep structures and measuring < 15 mm on diffusion-weighted (DWI) magnetic resonance imaging (MRI). Cortical strokes measuring <15 mm will qualify to be included in the study.
* Evidence of a cause explaining the stroke (e.g. hypercoagulable state or any other major source of cardiac embolism).

For TIA patients:

* Patients no fulfilling the criteria for ETUS.

For cerebral venous thrombosis patients:

* Subjects without involvement of the superior sagittal sinus (SSS)
* Subjects with an evident cause explaining the thrombosis (e.g., thrombophilia)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients with ESUS, ETUS, or SSS-CVTUS attending the Urgent TIA and Stroke Prevention Clinic or admitted to University or Victoria Hospital, in London, Ontario, Canada.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2025-03-29 (Estimated)

PRIMARY OUTCOMES:
Frequency of PNH in ESUS/ETUS/SSS-CVTUS | At recruitment
  Percentage of patients with flow-cytometry-confirmed PNH

SECONDARY OUTCOMES:
Frequency of PNH in ESUS/ETUS | At recruitment
  Percentage of ESUS/ETUS patients with flow-cytometry-confirmed PNH
Frequency of PNH in SSS-CVT | At recruitment
  Percentage of SSS-CVTUS patients with flow-cytometry-confirmed PNH

CONTACTS AND LOCATIONS:
Overall Officials: Luciano A Sposato, MD, Principal Investigator — London Health Sciences Center, Western University
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided